CLINICAL TRIAL: NCT00887315
Title: A Randomized Phase II Trial of Docetaxel, Cisplatin, and Hypofractionated Radiotherapy Versus Docetaxel and Cisplatin for Limited Volume Stage IV Non-small Cell Lung Cancer: The Synergistic Metastases Annihilation With Radiotherapy and Docetaxel (Taxotere) [SMART] Trial
Brief Title: The Synergistic Metastases Annihilation With Radiotherapy and Docetaxel (Taxotere) [SMART] Trial for Non-Small Cell Lung Cancer (NSCLC)
Acronym: SMART
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual and loss of sponsor
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16574B
Record Dates: First submitted 2009-04-22; First posted 2009-04-23 (Estimated); Results first posted 2013-12-06 (Estimated); Last update posted 2013-12-06 (Estimated); Status verified 2013-11

CONDITIONS: Non-small Cell Lung Cancer
Keywords: NSCLC; Metastatic Stage IV NSCLC; Limited Volume Stage IV Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Active Comparator): Chemotherapy only
  Interventions: Drug: Docetaxel and cisplatin
- 2 (Active Comparator): Chemotherapy and hypofractionated image guided radiotherapy
  Interventions: Radiation: Docetaxel and cisplatin Plus Hypofractionated Radiotherapy

INTERVENTIONS:
Drug: Docetaxel and cisplatin — Docetaxel 75 mg/m2 and cisplatin 75 mg/m2 IV repeated every 21 days for 2 additional cycles. For patients randomized to group 1, the chemotherapy is identical to that administered for the first 2 cycles
  Arms: Group 1
Radiation: Docetaxel and cisplatin Plus Hypofractionated Radiotherapy — Docetaxel 75 mg/m2 and cisplatin 75 mg/m2 IV for 2 cycles along with hypofractionated radiotherapy to all known sites of disease
  Arms: 2

SUMMARY:
Primary goal of the study is to assess the overall survival of the addition of hypofractionated image guided radiotherapy concurrently with Docetaxel and cisplatin. Survival will be assessed at 1 year from the date of study enrollment to date of death.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Life expectancy > 6 months
3. Histologically or cytologically confirmed diagnosis of NSCLC
4. Patients with AJCC stage IV cancer with distant metastases and without malignant pleural or pericardial effusion at diagnosis and before start of study

   1. Patients with pleural effusion that is transudative, cytologically negative, and non-bloody are eligible as long as they are stable and do not impair the ability to define tumor volumes.
   2. If a pleural effusion is too small for diagnostic thoracentesis, the patient will be eligible.
5. Primary and regional nodal disease that is encompassable in a reasonable radiotherapy portal:
6. Patients with 1-5 sites of disease and amenable to RT therapy as seen on standard imaging (CT, MRI, bone scan, PET scan)
7. Unidimensionally measurable disease (based on RECIST) is desirable but not strictly required.
8. Patients with brain metastases are allowed as long as they meet all other inclusion criteria. Brain metastases must be treated with whole brain radiotherapy and stereotactic radiosurgery or surgical resection followed by whole brain radiotherapy.
9. ECOG performance status <2
10. No prior RT to currently involved tumor sites
11. Baseline peripheral neuropathy < grade 1
12. Room air saturation (SaO2) > 90%
13. Patients must have normal organ and marrow function
14. Men and women of childbearing potential must be willing to consent to using effective contraception while on treatment and for at least 3 months thereafter.
15. Signed Informed consent
16. Inclusion of Women and Minorities
17. RT: Patient must have a completed treatment plan approved by the protocol review team

Exclusion Criteria:

1. Uncontrolled intercurrent illness including, but not limited to, ongoing active infection, symptomatic congestive heart failure (CHF), unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with the study requirements
2. Patients with clinically significant pulmonary dysfunction, cardiomyopathy, or any history of clinically significant CHF are excluded. The exclusion of patients with active coronary heart disease will be at the discretion of the attending physician.
3. Patients with significant atelectasis such that CT definition of the gross tumor volume (GTV) is difficult to determine.
4. < 1000 cc of tumor free lung.
5. Tumor volume and location which requires a lung volume-PTV >40% to receive >20 Gy (V20 <40%).
6. Patients with exudative, bloody, or cytologically malignant effusions are not eligible.
7. Pregnancy or breast feeding (Women of child-bearing potential are eligible, but must consent to using effective contraception during therapy and for at least 3 months after completing therapy)
8. Patients must have no uncontrolled active infection other than that not curable without treatment of their cancer.
9. Patients with a history of severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80.
10. Patient may not be receiving any other investigational agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-04; Primary Completion 2011-03 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Everett E Vokes, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Funding was withdrawn before conclusions were reached so the study was terminated.
Groups:
- Chemo Only: Chemotherapy only
- Chemo and Radiation: Chemotherapy and hypofractionated image guided radiotherapy
Period: Overall Study
Arm/Group | Chemo Only | Chemo and Radiation
Started | 7 | 4
Completed | 0 | 0
Not Completed | 7 | 4
Not completed — Study termination | 7 | 4

BASELINE CHARACTERISTICS:
Groups:
- Chemo and Radiation: Chemotherapy and radiotherapy
- Total: Total of all reporting groups
Arm/Group | Chemo Only | Chemo and Radiation | Total
Number analyzed (Participants) | 7 | 4 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 0 | 3
  >=65 years | 4 | 4 | 8
Age Continuous [Mean (Standard Deviation); unit: years] | 66.4 (10.6) | 74 (3.2) | 69.1 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: 1-Year Overall Survival
Description: Overall survival is assessed at 1 year from the date of study enrollment to date of death.
Time Frame: Baseline to death from any cause, 1 year
Population: The study was terminated before conclusions were reached so no data was analyzed.
Arm/Group | Chemo Only | Chemo and Radiation
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Overall PFS and CT Rate
Description: Overall PFS and CT rate is assessed response with PET and CT. Toxicity of addition of high dose focused RT to systemic therapy.Late (>90 day) radiotherapy toxicity will be assessed with RTOG/EORTC late RT toxicity guidelines
Time Frame: >90 days
Population: The study was terminated before conclusions were reached so no data was analyzed.
Arm/Group | Chemo Only | Chemo and Radiation
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: The adverse event data were not collected due to the study termination
Arm/Group | Chemo Only | Chemo and Radiation
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Funding was withdrawn before conclusions were reached so the study was terminated and no data was collected and analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No